CLINICAL TRIAL: NCT02790879
Title: Clinical Impact of the Transition From Pediatric to Adult Cystic Fibrosis Care Center
Brief Title: Transition From Pediatric to Adult Cystic Fibrosis Care Center
Acronym: SAFETIM RNM
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL15_0629
Record Dates: First submitted 2016-05-31; First posted 2016-06-06 (Estimated); Last update posted 2016-06-06 (Estimated); Status verified 2016-05

CONDITIONS: Cystic Fibrosis
Keywords: Transitional care; teenagers; cystic fibrosis; pulmonary function; nutritional function; Patients who experiment a transition pediatric - adult care
MeSH Terms: conditions — Cystic Fibrosis | interventions — Transition to Adult Care

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Transition: Patients who switched from pediatric cystic fibrosis care center to an adult cystic fibrosis care center during 2013 or 2014, regardless of their clinical status.
  Interventions: Other: Transition pediatric - adult

INTERVENTIONS:
Other: Transition pediatric - adult

SUMMARY:
The main objective of register-SAFETIM is to assess the impact of the transition from pediatric to adult cystic fibrosis care center on changes in lung function and nutritional status of patients.

This is a multicenter, observational, longitudinal, with analysis of the French national registry data of patients with cystic fibrosis.

Our study will assess the clinical features of adolescent patients with cystic fibrosis during the transition from pediatric care to adult care. It will explore factors associated with the impact of the transition on the clinical course of adolescent patients (respiratory and nutritional functions).

ELIGIBILITY:
Inclusion Criteria:

- patients who switched from pediatric cystic fibrosis care center to an adult cystic fibrosis care center during 2013 or 2014, regardless of their clinical status.

Exclusion Criteria:

- Patients whose transition year is not given in the French national register, that is to say patients from some mixed care center.

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients who switched from pediatric cystic fibrosis care center to an adult cystic fibrosis care center during 2013 or 2014, regardless of their clinical status
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2015-10; Primary Completion 2016-10 (Estimated); Study Completion 2016-10 (Estimated)

PRIMARY OUTCOMES:
Changes in FEV (FEV is the slope expressed in percentage of the predicted value). | Two years

SECONDARY OUTCOMES:
Body Mass Index (BMI) | Two years
Pseudomonas aeruginosa colonization | Two years
External pancreatic insufficiency | Two years
Diabetes | Two years

CONTACTS AND LOCATIONS:
Overall Officials: Sandrine TOUZET, MD, Principal Investigator — Hospices Civils de Lyon, Pôle Information Médicale, Evaluation, Recherche
Locations (1):
- Pôle Information Médicale, Evaluation, Recherche 162 avenue Lacassagne - Bâtiment A, Lyon, Auvergne-Rhône-Alpes, France